CLINICAL TRIAL: NCT01349491
Title: Ranolazine for the Prevention of Recurrent Persistent Atrial Fibrillation After Electrical Cardioversion: A Pilot Study
Brief Title: Ranolazine for the Prevention of Atrial Fibrillation After Electrical Cardioversion
Acronym: GILEAD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low recruitement rates
Sponsor: University of Oklahoma (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2399
Record Dates: First submitted 2011-04-25; First posted 2011-05-06 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Ranolazine
MeSH Terms: conditions — Atrial Fibrillation | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranolazine (Experimental): Patients will be started on ranolazine 500mg twice daily. The dose will be doubled after 2 weeks to 1000mg twice daily as tolerated.
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Patients will be started on a matching placebo twice daily. The first dose will be administered the day of cardioversion.
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Ranolazine — Patients will be started on ranolazine 500mg twice daily. The first dose will be administered the day of cardioversion. The dose will be doubled after 2 weeks to 1000mg twice daily as tolerated for a total of six months.
  Other Names: Ranexa
  Arms: Ranolazine
Drug: Matching placebo — Patients will be started on a matching placebo twice daily. The first dose will be administered the day of cardioversion and continued for a total of six months.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The investigators hypothesize that ranolazine would decrease the incidence of recurrence of Atrial Fibrillation (AF) after electrical cardioversion of persistent AF. Patients with persistent AF who are candidates for electrical cardioversion will be randomized to either placebo or ranolazine after successful electrical cardioversion.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common clinically significant cardiac arrhythmia and is associated with increased cardiovascular morbidity and mortality. Although a rhythm control strategy offers no survival benefit over a rate control strategy, elective electrical cardioversion is still recommended in patients without hemodynamic instability for symptomatic relief. However, recurrences are frequent after cardioversion and antiarrhythmic medications are required to maintain sinus rhythm. Nonetheless, the use of antiarrhythmic medications is problematic because of the risk of serious potential adverse effects, including drug-induced ventricular arrhythmias.

Ranolazine is a novel antianginal agent, which inhibits the late inward sodium current and produces antiischemic effects without reducing heart rate or blood pressure. Additionally, recent preclinical as well as preliminary clinical data suggest that ranolazine exhibits distinct antiarrhythmic properties. However, there is no controlled data for the use of ranolazine to prevent recurrence of AF after electrical cardioversion of persistent AF.

The investigators hypothesize that ranolazine would decrease the incidence of recurrence of AF after electrical cardioversion of persistent AF. Patients with persistent AF who are candidates for electrical cardioversion will be randomized to either placebo or ranolazine after successful electrical cardioversion. They will be followed at 2 weeks, 1, 3 and 6 months for clinical evaluation and electrocardiography for the detection of recurrence of AF.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with persistent atrial fibrillation, aged 21 or older
* Duration of atrial fibrillation less than one year
* The patient does not have any contraindications for anticoagulation
* The patient is willing to participate in the study for a total of 6 months with 3 outpatient office visits
* The patient has provided written informed consent during the screening visit to any test or procedure being performed, or medication being changed, for this study.
* The patient has no clinically significant abnormal clinical laboratory values, which in the investigator's opinion precludes the patient from safely participating in the study.

Exclusion Criteria:

* Any contraindication for anticoagulation
* New York Heart Association class IV heart failure
* Currently taking anti-arrhythmic drugs
* Chronic kidney disease (serum creatinine less than 2.5mg/dL) or severe liver dysfunction
* Pregnancy/nursing
* Prolonged QT interval (>500ms)
* Taking other medications known to prolong the QT interval
* Taking other medications known to affect the metabolism of ranolazine

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Udho Thadani, MD, Principal Investigator — University of Oklahoma; Stavros Stavrakis, MD, Study Director — University of Oklahoma
Locations (2):
- United States (2):
  - Oklahoma City VA Medical Center, Oklahoma City, Oklahoma
  - OU Medical Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ranolazine | Placebo
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome - Number of Participants With Atrial Fibrillation
Description: To determine if ranolazine is effective in decreasing recurrences of AF in patients with persistent AF successfully treated with electrical cardioversion.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 5 | 5
participants | 3 | 3

ADVERSE EVENTS:
Arm/Group | Ranolazine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No